CLINICAL TRIAL: NCT00078975
Title: A Phase II Study of Triapine in Combination With Gemcitabine in Recurrent/Unresectable/Metastatic Pancreatic Carcinoma
Brief Title: 3-AP and Gemcitabine in Treating Patients With Recurrent, Unresectable, or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMH-PHL-023; CDR0000353205 (Registry Identifier: PDQ (Physician Data Query)); NCI-6271
Record Dates: First submitted 2004-03-08; First posted 2004-03-09 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; recurrent pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

ARMS (1):
- Triapine in combination with Gemcitabine (Experimental)
  Interventions: Drug: gemcitabine hydrochloride; Drug: triapine

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: triapine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as 3-AP and gemcitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. 3-AP may help gemcitabine kill more tumor cells by making them more sensitive to the drug.

PURPOSE: This phase II trial is studying how well giving 3-AP together with gemcitabine works in treating patients with recurrent, unresectable, or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antitumor activity of 3-AP (Triapine®) and gemcitabine, in terms of complete and partial response and 6-month progression-free disease, in patients with recurrent, unresectable, or metastatic pancreatic cancer.

Secondary

* Determine the objective response rates, median survival, 1-year survival rate, duration of response or stable disease, and progression-free survival of patients treated with this regimen.
* Determine the safety and tolerability of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive 3-AP (Triapine®) IV over 2 hours and gemcitabine IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a complete or partial response receive an additional 2 courses of therapy beyond response.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 28-50 patients will be accrued for this study within 7-13 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed pancreatic adenocarcinoma

  * Recurrent, unresectable, or metastatic disease
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * Prior radiation field must not have encompassed the only site of measurable disease
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 12 weeks

Hematopoietic

* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No G6PD deficiency

Hepatic

* Bilirubin ≤ 1.5 times normal
* AST and ALT ≤ 2.5 times upper limit of normal

Renal

* Creatinine ≤ 1.5 times normal OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No unstable angina pectoris
* No cardiac arrhythmia
* No symptomatic congestive heart failure

Pulmonary

* No severe pulmonary disease
* No dyspnea at rest
* No dependence on supplemental oxygen use

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study treatment
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to study drugs
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other concurrent uncontrolled illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy except fluorouracil given as adjuvant therapy OR as a radiosensitizer during radiotherapy
* More than 4 weeks since prior adjuvant fluorouracil therapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* See Chemotherapy
* More than 4 weeks since prior radiotherapy and recovered

Surgery

* Not specified

Other

* No other concurrent investigational agents
* No other concurrent anticancer therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-04; Primary Completion 2005-12 (Actual); Study Completion 2009-01-07 (Actual)

PRIMARY OUTCOMES:
Objective response (complete and partial) | Every 8 weeks for the duration of the trial, an expected average of 5 years
Prolonged stable disease rate | Stable disease of 6 or more months

SECONDARY OUTCOMES:
Median survival | For duration of trial, an expected average of 5 years
Survival rate at 1 year | 1 year
Response duration | From date of response until progression
Progression-free survival | From date of response until progression or death
Safety and tolerability | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm J. Moore, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (4):
- Canada (4):
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario